CLINICAL TRIAL: NCT03965767
Title: Does The Combined Use Of Local And Intravenous Tranexamic Acid Offer Better Surgical Field Quality During Functional Endoscopic Sinus Surgery? A Placebo-Controlled Clinical Trial
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ossama Mustafa Mady, Ain Shams University, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FMASU R 27-2019
Record Dates: First submitted 2019-05-24; First posted 2019-05-29 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Chronic Sinus Disease; Nasal Polyps
Keywords: endoscopic sinus surgery- tranexamic acid
MeSH Terms: conditions — Nasal Polyps | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- control (Placebo Comparator)
  Interventions: Drug: Tranexamic Acid
- local group (Active Comparator)
  Interventions: Drug: Tranexamic Acid
- systemic group (Active Comparator)
  Interventions: Drug: Tranexamic Acid
- combined local and systemic (Active Comparator)
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Tranexamic Acid — comparison of effect of tranexamic acid on control of bleeding when used locally in the nose or systemic use

SUMMARY:
Functional Endoscopic Sinus surgery (FESS) is a surgery done for chronic rhinosinusitis after failure of medical treatment. Intraoperative bleeding poses a challenge to both the surgeon and anaesthetist. Although blood loss is not massive during FESS, bleeding may obscure the surgical field prolonging the time of surgery or even leading to incompletion of the surgery.

Different methods have been used to improve the surgical field but none without side effects. The use of diathermy carries the risk of local tissue damage with the risk of subsequent bleeding. Local vasoconstrictors carry the risk of systemic absorption. Induced hypotension may not be suitable for all patients; besides, this may necessitates the use of more anaestheic drugs with their associated side effects. In addition, none of theses methods have provided ideal surgical field for the surgeon.1-3 Tranexamic acid, an antifibrinolytic agent, has been used to decrease surgical field bleeding in different surgeries showing effectiveness in its topical, oral and intravenous use.4-6 The aim of this study is to evaluate the effectiveness of local, intravenous and combined use of tranexamic acid in improving the surgical field quality during functional endoscopic sinus surgery.

DETAILED DESCRIPTION:
After obtaining local ethical committee approval and written informed consent from the patients, 90 adult patients of both sex, aged between 18 and 50 years, ASA I-II, scheduled for elective functional endoscopic sinus surgery in Ain Shams University hospitals will be enrolled in this randomized, controlled prospective double blinded study.

Exclusion criteria included; patients with uncontrolled hypertension or coronary artery disease, anaemia, end stage renal failure, liver cirrhosis, patients with coagulopathy or receiving drugs influencing blood coagulation, cerebrovascular thrombosis or history of thrombotic events, pregnancy, known sensitivity to any of the study drug and patients' refusal to participate in the study.

The surgeon will assess the degree of sinus involvement in each patient using the Lund-Mackay scoring system. All the patients will be instructed to take prednisone 1 mg. kg-1 5 days before surgery to reduce inflammation.

After applying basic monitors, all patients will be premedicated with midazolam 0.05 mg.kg -1 IV, ranitidine 50 mg IV and dexamethasone 10 mg IV, 15 min. prior to surgery.

In the operating room and after 5 min preoxygenation, general anesthesia will be conducted using the same protocol for all patients: fentanyl 1 μg.Kg-1, propofol 2-2.5 mg.kg -1 and atracurium 0.5 mg. Kg-1 to facilitate endotracheal intubation.

Anaesthesia will be maintained using isoflurane 1 -1.5% in oxygen and air mixture 1:1 and atracurium 0.1 mg. Kg-1 every 30 mim. Positive pressure ventilation was set to maintain normocapnia. Fentanyl bolus of 0.5 μg.Kg-1 to maintain MAP (60-70 mmHg), without exceeding a total dose of 5 μg.Kg-1 for fast tracking and early extubation. Total dose of fentanyl will be recorded.

A throat pack soaked with saline will be inserted in all patients to prevent blood from reaching the gastrointestinal track. The surgeon will insert nasal pack (epinephrine 1/2000 soaked pack), Afterwards, he will inject 2 ml of epinephrine 1:100000 into the middle turbinate and the junction of the middle turbinate to the lateral nasal wall. All patients will be placed in the same position.

Patients will then be randomly and evenly assigned to one of the four groups, 30 patients each.

Group I: patients will receive an intravenous dose of 15 mg.kg-1 of tranexamic acid in a 10 ml syringe. The irrigation fluid will be 400 ml of normal saline.

Group II: patients will receive intravenous dose of 10 ml normal saline in 10 ml syringe. Irrigation fluid will be 400 ml of normal saline with 2 g of tranexamic acid added to it. If more irrigation is needed, normal saline will be used.

Group III: patients will receive an intravenous dose of 15 mg.kg-1 of tranexamic acid in a 10 ml syringe. Irrigation fluid will be 400 ml of normal saline with 2 g of tranexamic acid added to it. If more irrigation is needed, normal saline will be used.

Group IV (control): patients will receive intravenous dose of 10 ml normal saline in 10 ml syringe. The irrigation fluid will be 400 ml of normal saline.

Randomization was done using computer generated list. A pharmacist will prepare the drugs, as well as the irrigation fluid, which will only have the patient's number on them. In this way, the anaesthetist and the surgeon will be blinded to the study groups. The same surgeon performed all the operations.

In all groups, if bleeding was uncontrollable and affecting the surgical field, loading dose of esmolol 500 μg.Kg-1 will be started, followed by infusion of 100-300 mg.Kg-1.min-1. The use and total dose of esmolol will be reported.

MAP and HR will recorded before induction of anaesthesia (baseline), immediately after induction, and every 15 mim till completion of surgery.

Beside the maintenance fluid infusion, intraoperative blood loss will be compensated with crystalloids in a ratio of 1:3.

Prothrombin time (PT), partial thromboplastin time (PTT) and complete blood count (CBC) will be measured before surgery and 6 hours after surgery.

The surgeon will be asked to estimate the surgical field on a 5-point Boezaart scale immediately at the end of the surgery (table 1).

Table 1: Surgical field quality based on Boezaart scale. 7 Grade Assessment 0 No bleeding.

1. Slight bleeding, no suction of blood required.
2. Slight bleeding, occasional suction required.
3. Slight bleeding, frequent suction required. Bleeding threatens surgical field few seconds after suction is removed.
4. Moderate bleeding, frequent suction required. Bleeding threatens surgical field directly after suction is removed.
5. Severe bleeding, constant suction required. Bleeding appears faster than can be removed by suction. Surgical field severely threatened and surgery not possible

The incidence of postoperative complications including; epistaxis, nausea, vomiting and pain (using VAS) will be evaluated in the PACU.

ELIGIBILITY:
Inclusion Criteria:

* patients underwent endoscopic sinus surgery

Exclusion Criteria:

* patients with uncontrolled hypertension or coronary artery disease, anaemia, end stage renal failure, liver cirrhosis, patients with coagulopathy or receiving drugs influencing blood coagulation, cerebrovascular thrombosis or history of thrombotic events, pregnancy, known sensitivity to any of the study drug and patients' refusal to participate in the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-04-25 (Actual); Primary Completion 2019-08-25 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
bleeding during surgery | time of surgery
  surgeon satisfaction

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Ain Shams University, Cairo, Egypt